CLINICAL TRIAL: NCT00005444
Title: Hypertension in Families of African Origin
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4373; R29HL052075 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2004-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To investigate familial patterns of hypertension and related cardiovascular (CV) risk factors in the United States and Nigeria.

DETAILED DESCRIPTION:
BACKGROUND:

It has been known for many years that African Americans experience twofold higher rates of hypertension than do whites. The underlying biological mechanisms which lead to this differential are still not understood, however. Despite widespread speculation that persons of African descent are genetically susceptible to hypertension, few direct studies have been carried out. Rates of hypertension remain low in West Africa, and this study will provide a contrast between populations of similar genetic background in a low versus high risk environmental setting

DESIGN NARRATIVE:

A total of 240 families were identified from completed community surveys in Maywood, Illinois and Ibadan, Nigeria. Probands were ages 45-55 and equally divided between males and females. A minimum of five first-degree relatives were examined in each family to obtain information on the following variables: blood pressure (BP), obesity, urinary sodium and potassium, socioeconomic status and physical activity. In addition, plasma and DNA were collected and stored for future studies of relevant physiologic intermediate phenotypes and candidate genes for hypertension in the two contrasting populations. These data provided the basis for examining familial aggregation of blood pressure/hypertension and related CV risk factors. Three primary goals were addressed: 1) to determine whether the familial aggregation of blood pressure in Black populations was influenced by the overall distribution of environmental factors at the population level, by contrasting the distribution of familial correlations of blood pressure and the familial aggregation of hypertension, in Nigeria and the United States; to determine the significance of measured environmental correlates of blood pressure by comparing the magnitude of variance components for probands and relatives in each setting; and 3) to use path analysis to obtain estimates of genetic and cultural heritability of blood pressure, controlling for clustering environmental factors at the household level. Plasma and DNA samples collected in this study provided additional valuable resources for future molecular research.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-08; Study Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Rotimi — Howard University

REFERENCES:
- [Background] Rotimi C, Luke A, Li Z, Compton J, Bowsher R, Cooper R. Heritability of plasma leptin in a population sample of African-American families. Genet Epidemiol. 1997;14(3):255-63. doi: 10.1002/(SICI)1098-2272(1997)14:33.0.CO;2-4. PMID 9181355
- [Background] Rotimi C, Cooper R, Ogunbiyi O, Morrison L, Ladipo M, Tewksbury D, Ward R. Hypertension, serum angiotensinogen, and molecular variants of the angiotensinogen gene among Nigerians. Circulation. 1997 May 20;95(10):2348-50. doi: 10.1161/01.cir.95.10.2348. PMID 9170394
- [Background] Rotimi CN, Cooper RS, Cao G, Ogunbiyi O, Ladipo M, Owoaje E, Ward R. Maximum-likelihood generalized heritability estimate for blood pressure in Nigerian families. Hypertension. 1999 Mar;33(3):874-8. doi: 10.1161/01.hyp.33.3.874. PMID 10082502
- [Background] Rotimi CN, Comuzzie AG, Lowe WL, Luke A, Blangero J, Cooper RS. The quantitative trait locus on chromosome 2 for serum leptin levels is confirmed in African-Americans. Diabetes. 1999 Mar;48(3):643-4. doi: 10.2337/diabetes.48.3.643. No abstract available. PMID 10078570
- [Background] Luke A, Rotimi CN, Adeyemo AA, Durazo-Arvizu RA, Prewitt TE, Moragne-Kayser L, Harders R, Cooper RS. Comparability of resting energy expenditure in Nigerians and U.S. blacks. Obes Res. 2000 Aug;8(5):351-9. doi: 10.1038/oby.2000.42. PMID 10968726
- [Background] Okosun IS, Liao Y, Rotimi CN, Prewitt TE, Cooper RS. Abdominal adiposity and clustering of multiple metabolic syndrome in White, Black and Hispanic americans. Ann Epidemiol. 2000 Jul;10(5):263-70. doi: 10.1016/s1047-2797(00)00045-4. PMID 10942873
- [Background] Schork NJ, Chakravarti A, Thiel B, Fornage M, Jacob HJ, Cai R, Rotimi CN, Cooper RS, Weder AB. Lack of association between a biallelic polymorphism in the adducin gene and blood pressure in whites and African Americans. Am J Hypertens. 2000 Jun;13(6 Pt 1):693-8. doi: 10.1016/s0895-7061(00)00237-5. PMID 10912755
- [Background] Cooper RS, Guo X, Rotimi CN, Luke A, Ward R, Adeyemo A, Danilov SM. Heritability of angiotensin-converting enzyme and angiotensinogen: A comparison of US blacks and Nigerians. Hypertension. 2000 May;35(5):1141-7. doi: 10.1161/01.hyp.35.5.1141. PMID 10818078
- [Background] Colilla S, Rotimi C, Cooper R, Goldberg J, Cox N. Genetic inheritance of body mass index in African-American and African families. Genet Epidemiol. 2000 Apr;18(4):360-76. doi: 10.1002/(SICI)1098-2272(200004)18:43.0.CO;2-H. PMID 10797595